CLINICAL TRIAL: NCT04207697
Title: Study to Assess the Safety and Effectiveness of Beltavac® Polymerized With Cat Dander
Status: Completed | Type: Observational
Sponsor: Probelte Pharma S.L.U. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-BEL-2019-01
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Rhinoconjunctivitis With or Without Allergic Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Beltavac® Polymerized with cat dander — Adminstration of Beltavac® Polymerized with cat dander according to the routine clinical practice

SUMMARY:
Non-interventional Study to Assess the Safety and Effectiveness Profile of a SCIT Therapy With Beltavac® Polymerized With Cat Dander in allergic patients

DETAILED DESCRIPTION:
This prospective open multi-centre non-interventional study assess the safety and effectiveness profile of the subcutaneous allergen-specific immunotherapy with Beltavac® Polymerized with cat dander allergic patients (children and adults) in routine medical care. Patients receive a rush schedule administration every month for a year. They attend at least 5 study visits to inform about the adverse reactions, the self reported symptoms and the medication intake.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the age of 12 years and older suffering from a clinically relevant cat dander induced allergic rhinitis or rhinoconjunctivitis associated with or not with asthma
* Positive skin testing
* Positive Serum-Specific IgE determination
* Informed consent

Exclusion Criteria:

* Patients suffering from acute or chronic infections or inflammations
* Patients suffering from uncontrolled asthma
* Patients with a known autoimmune disease
* Patients with active malignant disease
* Patients requiring beta-blockers
* Patients having any contraindication for the use of adrenaline
* Patients with previous immunotherapy with this allergen or another allergen with cross-reaction
* Patients with immunotherapy treatment at the time of inclusion

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 12 years or older who suffer from allergic rhinoconjunctivitis caused by cat dander
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Numbers of treatment-related local and systemic reactions | 12 months
  Number of adverse reactions occurred during the treatment period and classified according to the WAO standards

SECONDARY OUTCOMES:
Combined Symptom and Medication Score of Rhinoconjunctivitis | 12 months
  The score will be calculated as a sum of the symptoms score (0-3) and medication score (0-3)
Combined Symptom and Medication Score of Asthma | 12 months
  The score will be calculated as a sum of the symptoms score (0-3) and medication score (0-3)
Visual analogue Scale Score | 12 months
  Psycometric scale that assesses the global allergic disease discomfort. It is a 10 cm line representing severity from 0:"no symptoms" to 10 "highest level of symptoms"
IgE and IgG4 specific quantification | 6 and 12 months
  IgE and IgG4 quantification in serum at baseline, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Mérida, Principal Investigator — San Cecilio Universitary Hospital
Locations (7):
- Spain (7):
  - Campus de la Salud University Hospital, Granada, Andalusia
  - Ciudad de Jaen Hospital, Jaén, Andalusia
  - Quirón Campo de Gibraltar Hospital, Palmones, Cádiz
  - Quirón Malaga Hospital, Málaga, Malaga
  - Al-lergo Centre Clinic, Barcelona
  - Bellvitge University Hospital, Barcelona
  - Alergogranada, Granada